CLINICAL TRIAL: NCT00723671
Title: Magnetic Resonance Spectroscopy, Perfusion and Diffusion Tensor Imaging in Neuropsychiatric Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Pia C Maly Sundgren, MD, PhD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00050562
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Systemic Lupus Erythematosus; Fibromyalgia; Acute Neuropsychiatric Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fibromyalgia

ARMS (1):
- metabolic peaks (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI

SUMMARY:
The purpose of this study is to find out if certain types of Magnetic Resonance (MR) scanning will help to better detect markers in the brain that are related to the neuropsychiatric symptoms of systemic lupus erythematosus (SLE). A small percentage of patients who have this type of lupus experience symptoms that may result from a blood clot or change in blood vessel structure in the brain. These neuropsychiatric symptoms can include an inability to think clearly, a change in level of awake and/or awareness, and in the worst cases, seizure and stroke. Another goal of the study is to find out if individuals with fibromyalgia (FM), or chronic pain, have symptom-related markers in any of these scans as well. Better and earlier detection of markers that are related to acute neuropsychiatric lupus (NPSLE) and FM will be helpful to all who are affected by these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology (ACR) criteria for SLE with neuropsychiatric symptoms.
* Be 18 years of age or older.
* Have recent onset of neurological symptoms that have been active within the last 14 days. The criteria for NPSLE study patients will be a clinically significant neurologic examination which, in the opinion of the treating physician, may be due to SLE and requires MRI evaluation. Patients will be classified according to the nomenclature recommended by the ACR on Neuropsychiatric Manifestations in SLE, and further classified as "focal," "nonfocal," or "seizure" [68].
* Be willing and able to complete all study procedures and sign the informed consent form.
* Report no neurological symptoms at the time of enrollment.
* The patients meeting the baseline criteria will be sequentially enrolled from the Lupus Cohort. Recruitment will be adjusted to include equal numbers of APA positive and APA negative patients.
* Meet the established ACR criteria for FM [69].
* Be willing and able to complete all study procedures associated with baseline scanning.

Exclusion Criteria:

* Those SLE patients with acute onset of neurological symptoms with duration longer than 14 days.
* Individuals who are pregnant.
* Individuals who are left-handed.
* Individuals who meet 1990 ACR criteria for FM
* Have acute onset of neurological symptoms related to SLE.
* Individuals who are pregnant.
* Individuals who are left-handed.
* Individuals who meet ACR criteria for FM.
* Co-morbid medical illnesses capable of causing a worsening of physical functional status independent of the diagnosis (e.g., morbid obesity), autoimmune diseases other than SLE cardiopulmonary disorders (e.g., angina, congestive heart failure, COPD(chronic obstructive pulmonary disease), chronic asthma), uncontrolled endocrine or allergic disorders (e.g., thyroid dysfunction, Type I diabetes), and malignancy within 2 years, excluding successfully treated squamous or basal skin carcinoma.
* Any present psychiatric disorder involving a history of psychosis (e.g., schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, etc.), current suicide risk or attempt within 2 years of the study, or substance abuse within 2 years.
* Individuals with mood disorders will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-11; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
differences in NAA | years

CONTACTS AND LOCATIONS:
Overall Officials: Pia Maly-Sundgren, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States